CLINICAL TRIAL: NCT03765879
Title: Brain Mechanisms of Video-Guided Acupuncture Imagery Treatment on Chronic Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018P002553
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: In this study, participants will be randomly assigned to receive one of two interventions: verum video-guided acupuncture imagery treatment (VGAIT) or sham VGAIT.
Who Masked: Investigator, Outcomes Assessor
Masking Description: This experiment will not be blinded. Participants will be aware if they are in the verum VGAIT or sham VGAIT group by nature of the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum VGAIT Group (Experimental): Participants in this group will receive verum (real) acupuncture and verum video-guided acupuncture imagery treatment (VGAIT).
  Interventions: Other: Verum VGAIT (Video-Guided Acupuncture Imagery Treatment)
- Sham VGAIT Group (Placebo Comparator): Participants in this group will receive sham acupuncture and sham VGAIT.
  Interventions: Other: Sham VGAIT (Video-Guided Acupuncture Imagery Treatment)

INTERVENTIONS:
Other: Verum VGAIT (Video-Guided Acupuncture Imagery Treatment) — In VGAIT treatment sessions, participants will re-watch the video of an avatar receiving acupuncture treatment, and they will be asked to vividly imagine that the treatment is being concurrently applied on themself.
  Arms: Verum VGAIT Group
Other: Sham VGAIT (Video-Guided Acupuncture Imagery Treatment) — In sham VGAIT treatment sessions, participants will re-watch this video of an avatar receiving the sham acupuncture treatment, and they will be asked to vividly imagine that the treatment is being concurrently applied on themself.
  Arms: Sham VGAIT Group

SUMMARY:
In this study, the investigators will examine the analgesic effects of acupuncture imagery treatment in patients with chronic low back pain. The intervention used in this study is "video-guided acupuncture imagery treatment" (VGAIT) treatment. The control used in this study is sham (fake) VGAIT. Participants in each group will participate in 8 study sessions (including 6 treatment sessions) over the course of 6 weeks. The primary outcome measure for this study is change in low back pain severity score after each treatment session.

DETAILED DESCRIPTION:
Low back pain is the one of the most common reasons for all physician visits in the USA and a leading cause of disability. However, conventional/pharmacological treatments for chronic low back pain (cLBP) have achieved limited success. Imagery is a commonly used therapeutic method for many disorders, such as chronic pain and stroke. Yet, the underlying mechanism remains unclear. Studies suggest that in addition to directly perceiving one's environment, individuals spend considerable time recalling and/or imagining experiences. A large body of literature suggests that common brain areas are activated during direct and vicarious (observational) experiences. Acupuncture is an invasive treatment that involves needle insertion and manipulation. Literature suggests that deqi (sensations evoked by acupuncture needle manipulation, such as soreness, aching, and dull pain) are crucial for treatment effects. In a recent study, the investigators examined video-guided acupuncture imagery treatment ("VGAIT"), during which participants watch a video of acupuncture previously administered on their own body while imagining it being concurrently applied. They found that this treatment can produce deqi sensations and increase pain thresholds in healthy subjects. In this study, the investigators will further investigate the modulation effects of VGAIT on patients with chronic pain.

This study will recruit up to 80 male and female participants, ages 18-60, with a diagnosis of chronic low back pain (having low back pain for more than 6 months), until 60 participants have finished the study. These participants will be randomly assigned to receive VGAIT or sham VGAIT, with 30 in each group.

We first performed a pilot study in which subjects (up to 25) only received real treatment to ensure that the intervention has a treatment effect. In addition, we will also compare the results from the pilot study with previous acupuncture studies from our lab to further validate the effect of VGAIT. If a treatment effect is evident in this pilot cohort, we will begin randomization.

This study consists of 10 sessions over approximately 6 weeks. These sessions include 2 assessment sessions (Session 1 and 10) and 8 treatment sessions (Sessions 2-9). The treatment sessions will consist of verum VGAIT or sham VGAIT. Verum VGAIT will involve the use of acupuncture points commonly used for chronic low back pain. Sham VGAIT will involve the use of non-acupoints.

All study procedures will take place in the department of Psychiatry or the Clinical Research Center at the Martinos Center for Biomedical Imaging (Charlestown Navy Yard Campus of Massachusetts General Hospital).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers 18-60 years of age
* Meet the Classification Criteria of the chronic low back pain (having low back pain for more than 6 months), as determined by the referring physician.
* At least 4/10 clinical pain on the 11-point low back pain intensity scale.
* Must have had a prior evaluation of their low back pain by a health care provider, which may have included radiographic studies. Documentation of this evaluation will be sought from Partners or outside medical records and kept in the subject's research record.
* At least a 10th grade English-reading level; English can be a second language provided that the patients feel they understand all the questions used in the assessment measures.

Exclusion Criteria:

* Specific causes of back pain (e.g. cancer, fractures, infections),
* Complicated back problems (e.g. prior back surgery, medico legal issues),
* Possible contraindications for acupuncture (e.g. coagulation disorders, cardiac pacemakers, pregnancy, seizure disorder), and conditions that might confound longitudinal effects or interpretation of results (e.g. severe fibromyalgia, rheumatoid arthritis).
* Conditions making study participation difficult (eg, paralysis, psychoses, or other severe psychological problems as per the judgment of a study investigator during Session 1)
* The intent to undergo surgery during the time of involvement in the study.
* History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome. For example: asthma or claustrophobia.
* Unresolved medical legal/disability/workers compensation claims in connection with low back pain.
* Active substance abuse disorder in the past 24 months, as determined by self-report and/or urine toxicology
* Lacking the capacity to consent for oneself

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in low back pain (LBP) severity score | 6 weeks
  LBP Severity will be measured by a single-item questionnaire that asks participants to rate how bothersome their back pain has been during the past week on a visual analog scale.

SECONDARY OUTCOMES:
Changes in back-pain specific disability score | 6 weeks
  Back-pain specific disability will be measured via the Roland-Morris Disability Questionnaire, an instrument that asks participants to describe their low back pain by using 24 questions. Higher scores on this instrument indicate more severe disability.
Changes in dysfunction, as measured by Patient Reported Outcomes Measurement System-29 (PROMIS-29) score | 6 weeks
  PROMIS-29 is a 29-item instrument that assesses pain, function, anxiety, and depression. Higher scores can indicate better or worse outcomes, depending on the section of this instrument being scored.
Changes in dysfunction, as measured by Patient Reported Outcomes Measurement System (PROMIS) Global Health score | 6 weeks
  PROMIS Global Health is a 10-item instrument that assesses pain, function, depression, and anxiety. A higher score on this instrument is associated with more improved outcomes in regard to these measures.
Changes in psychiatric symptoms as measured by PROMIS-29 | 6 weeks
  PROMIS-29 is a 29-item instrument that assesses pain, function, anxiety, and depression. Higher scores can indicate better or worse outcomes, depending on the section of this instrument being scored.
Changes in psychiatric symptoms as measured by PROMIS Global Health | 6 weeks
  PROMIS Global Health is a 10-item instrument that assesses pain, function, depression, and anxiety. A higher score on this instrument is associated with more improved outcomes in regard to these measures.
Changes in psychiatric symptoms as measured by Beck Depression Inventory (BDI-II) | 6 weeks
  BDI-II is a 210item instrument that is used to measure major depression. Higher scores on this instrument indicate more severe depression symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

REFERENCES:
- [Derived] Hodges S, Li Y, Wu J, Ma L, Liu Y, Reddy S, Sacca V, Walker KM, Chen L, Camprodon JA, Orr SP, Fregni F, Zhang Y, Yao S, Vangel M, Kong J. Novel avatar-based video-guided acupuncture imagery treatment for chronic low back pain: a randomised controlled trial in the USA. EClinicalMedicine. 2025 Oct 10;89:103538. doi: 10.1016/j.eclinm.2025.103538. eCollection 2025 Nov. PMID 41140457